CLINICAL TRIAL: NCT04132505
Title: Binimetinib Plus Hydroxychloroquine in KRAS Mutant Metastatic Pancreatic Cancer
Brief Title: Binimetinib and Hydroxychloroquine in Treating Patients With KRAS Mutant Metastatic Pancreatic Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-0191; NCI-2019-04991 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-0191 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-08-22; First posted 2019-10-18 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Metastatic Pancreatic Adenocarcinoma; Stage IV Pancreatic Cancer AJCC v8
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — binimetinib; Hydroxychloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (binimetinib, hydroxychloroquine) (Experimental): Patients receive binimetinib PO BID and hydroxychloroquine PO BID on days 1-14. Cycles repeat every 14 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Binimetinib; Drug: Hydroxychloroquine

INTERVENTIONS:
Drug: Binimetinib — Given PO
  Other Names: ARRY-162; ARRY-438162; MEK162; Mektovi
Drug: Hydroxychloroquine — Given PO

SUMMARY:
This phase I trial studies the best dose of hydroxychloroquine when given together with binimetinib in treating patients with KRAS gene mutated pancreatic cancer that has spread to other places in the body (metastatic). Binimetinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Hydroxychloroquine may prevent autophagy, a normal process in which a cell destroys proteins and other substances which may lead to cell death. Autophagy may prevent normal cells from developing into tumor cells, but it may also protect tumor cells by destroying anticancer drugs or substances taken up by them. Giving hydroxychloroquine together with binimetinib may work better in treating patients with pancreatic cancer compared to binimetinib alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the maximum tolerated dose of hydroxychloroquine (HCQ) when combined with a fixed dose of binimetinib.

SECONDARY OBJECTIVES:

I. To determine the response rate among a pilot cohort of pancreatic cancer patients.

II. To determine the safety and toxicity profile of the combination of binimetinib and HCQ.

III. To determine the ability of the combination to halt tumor growth as measured by progression free survival.

IV. To assess the overall survival of patients treated on this regimen.

EXPLORATORY OBJECTIVES:

I. To compare the efficacy of treatment to somatic gene mutation profile as acquired by standard of care testing.

II. To assess pre- and post- treatment tissue to determine if markers of autophagy correlate with response to treatment.

III. To assess the effect of this binimetinib/HCQ treatment on changes in muscle and fat mass as analyzed by computed tomography (CT) scan (as standard of care treatment).

OUTLINE: This is a dose-escalation study of hydroxychloroquine.

Patients receive binimetinib orally (PO) twice daily (BID) and hydroxychloroquine PO BID on days 1-14. Cycles repeat every 14 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Have histologically or cytologically confirmed diagnosis of pancreatic adenocarcinoma based on pathology report with radiologically identified metastases that meet Response Evaluation Criteria in Solid Tumors (RECIST) criteria.
* Be willing and able to provide written informed consent for the trial.
* Have at least one measurable lesion by RECIST criteria.
* Have had prior treatment with at least one line of therapy for metastatic disease.
* Have had tumor mutation profiling from any Clinical Laboratory Improvement Act (CLIA) certified laboratory demonstrating a KRAS mutation. Liquid biopsy demonstrating KRAS mutation will be considered acceptable.
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) performance scale.
* Absolute neutrophil count (ANC) >= 1500/uL (specimens must be collected within 10 days prior to the start of trial treatment).
* Platelets >= 100,000/uL (specimens must be collected within 10 days prior to the start of trial treatment).
* Hemoglobin >= 9.0 g/dL (specimens must be collected within 10 days prior to the start of trial treatment).
* Creatinine OR measured or calculated creatinine clearance (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl]) =< 1.5 x upper limit of normal (ULN) OR >= 50 mL/min for subjects with creatinine level > 1.5 x ULN (specimens must be collected within 10 days prior to the start of trial treatment).
* Total bilirubin =< 1.5 x ULN (specimens must be collected within 10 days prior to the start of trial treatment).
* Indirect bilirubin =< ULN (specimens must be collected within 10 days prior to the start of trial treatment).
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]), and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x ULN (=< 5 x ULN for subjects with liver metastases) (specimens must be collected within 10 days prior to the start of trial treatment).
* Alkaline phosphatase =< 2.5 x ULN (=< 5 x ULN for subjects with liver metastases) (specimens must be collected within 10 days prior to the start of trial treatment).
* Serum albumin > 3.3 mg/dl (specimens must be collected within 10 days prior to the start of trial treatment).
* International normalized ratio (INR) OR prothrombin time (PT), activated partial thromboplastin time (aPTT) =< 1.5 x ULN unless subject is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants (specimens must be collected within 10 days prior to the start of trial treatment).
* Female subjects of childbearing potential must have a negative urine or serum pregnancy test prior to the start of treatment.
* The participant is deemed by the investigator to have the ability to be compliant with scheduled visits, treatment plan, and study procedures.
* Male and female subjects of childbearing potential must agree to use an adequate method of contraception starting with the first dose of trial therapy through 30 days after the last dose of trial therapy. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject. Acceptable methods of contraception are listed in the protocol text.

Exclusion Criteria:

* Has pancreatic tumor other than adenocarcinoma, including: acinar cell carcinoma, pancreaticoblastoma, malignant cystic neoplasms, endocrine neoplasms, squamous cell carcinoma, ampulla of Vater, periampullary, duodenal, or common bile duct malignancies. Poorly differentiated carcinoma may be included at the discretion of the investigator if histologic features suggest the possibility of adenocarcinoma.
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational treatment within 2 weeks prior to the anticipated first dose of study treatment.
* Received anticancer therapy including chemotherapy, immunotherapy, or antineoplastic biologic drugs (e.g. erlotinib) within 14 days of the anticipated start of study treatment.
* Have undergone major surgery (e.g. inpatient procedures) =< 6 weeks prior to the start of study treatment or who have not recovered from side effects of earlier such procedures.
* Have undergone radiation within 7 days prior to the start of treatment.
* Patient has not recovered to =< grade 1 from toxic effects of prior therapy before starting study treatment. Note that alopecia, neuropathy, myalgias, and endocrinopathy are exceptions to this criteria.
* Impaired cardiovascular function or clinically significant cardiovascular disease including, but not limited to, any of the following:

  * History of acute coronary syndromes (including myocardial infarction, unstable angina, coronary artery bypass grafting, coronary angioplasty or stenting) < 6 months prior to screening;
  * Congestive heart failure requiring treatment (New York Heart Association grade >= 2);
  * Left ventricular ejection fraction (LVEF) < 50% as determined by multigated acquisition scan (MUGA) or echocardiography (ECHO);
  * Uncontrolled hypertension defined as persistent systolic blood pressure >= 150 mmHg or diastolic blood pressure >= 100 mmHg despite current therapy;
  * History or presence of clinically significant cardiac arrhythmias (including resting bradycardia, uncontrolled atrial fibrillation or uncontrolled paroxysmal supraventricular tachycardia);
  * Triplicate average baseline corrected QT (QTc) interval >= 480 ms.
* Impairment of gastrointestinal function or disease which may significantly alter the absorption of study drug (e.g., active ulcerative disease, uncontrolled vomiting or diarrhea, malabsorption syndrome, small bowel resection with decreased intestinal absorption), or recent (=< 3 months) history of a partial or complete bowel obstruction, or other conditions that will interfere significantly with the absorption of oral drugs.
* Had a solid organ or hematologic transplant.
* Concurrent neuromuscular disorder that is associated with elevated creatine kinase (CK) (e.g., inflammatory myopathies, muscular dystrophy, amyotrophic lateral sclerosis, spinal muscular atrophy).
* Has required treatment for other malignancies within 1 year prior to first dose of study treatment, with the exception of curatively treated basal cell carcinoma of the skin, squamous cell carcinoma of the skin and/or curatively resected tumors of low invasive potential (e.g., in situ cervical and/or breast cancers).
* Has a history of central nervous system (CNS) metastases and/or carcinomatous meningitis.
* History or current evidence of retinal vein occlusion (RVO) or current risk factors for RVO (e.g., uncontrolled glaucoma or ocular hypertension, history of hyperviscosity or hypercoagulability syndromes); history of retinal degenerative disease.
* Has an active infection requiring systemic therapy.
* Chronic use of steroids for pain or emesis management.
* Has known ophthalmologic disease that, in the opinion of investigators, would pose an increased risk of visual disturbances during the study. This includes a history or current evidence of retinal vein occlusion (RVO) or current risk factors for RVO (e.g., uncontrolled glaucoma or ocular hypertension, history of hyperviscosity or hypercoagulability syndromes); history of retinal degenerative disease. The routine use of eyeglasses does not in itself disqualify patient participation.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 30 days after the last dose of trial treatment.
* Has a known history of human immunodeficiency virus (HIV) infection (HIV 1/2 antibodies) (No HIV screening is required for patients with no known diagnosis).
* Has a history of the following liver diseases:

  * Hepatitis B (defined as hepatitis B surface antigen [HBsAg] reactive),
  * Hepatitis C (defined as detectable hepatitis C virus [HCV] ribonucleic acid [RNA]),
  * Primary biliary cholangitis,
  * Primary sclerosing cholangitis,
  * History of immune mediated cholangitis.
  * Of note, patients with a history of bacterial cholangitis are eligible if the infection has been fully resolved prior to the screening visit. An exception is made for hepatitis C patients who have undergone treatment and who have negative serologic testing for at least one year.
* Has a known history of active TB (Mycobacterium Tuberculosis).
* Is unable to tolerate a contrast enhanced computed tomography (CT) or magnetic resonance imaging (MRI) for staging/restaging purposes.
* In the estimation of the treating physician or primary investigator, have had a clinical deterioration of their ECOG performance within the month prior to enrollment. Evidence for such deterioration shall be documented in the patient's medical record.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator. Evidence for such abnormalities/conditions will be documented in the patient's medical record.
* Has a history of thromboembolic or cerebrovascular events =< 12 weeks prior to the first dose of study treatment. Examples include transient ischemic attacks, cerebrovascular accidents, hemodynamically significant (i.e. massive or sub-massive) deep vein thrombosis or pulmonary emboli. Note: Patients with either deep vein thrombosis or pulmonary emboli that does not result in hemodynamic instability are allowed to enroll as long as they are on a stable dose of anticoagulants for at least 4 weeks. Also note: Patients with thromboembolic events related to indwelling catheters or other procedures may be enrolled. Finally: patients with stable mesenteric thrombosis that predate study assessment (eg portal vein thrombus) may be enrolled.
* Has a history of active bleeding requiring transfusion within a 3 month period prior to screening. (Transfusions attributed to chemotherapy related anemia do not meet this exclusion criterion.)
* Known cases of drug-induced hepatobiliary toxicities (other than a radiological finding of fatty liver).
* Has had prior treatment with a MEK or ERK inhibitor.
* Partial or complete bowel obstruction.
* Impaired gastrointestinal function that may significantly alter the absorption of binimetinib (e.g., ulcerative diseases, uncontrolled vomiting, malabsorption syndrome, small bowel resection with decreased intestinal absorption) or baseline diarrhea >= grade 1.
* Use of digoxin, mefloquine, cyclosporine, methotrexate, fexofenadine, quinidine, talinolol, vinblastine, coumestrol, daidzein, dantrolene, estrone-3-sulfate, genistein, prazosin, sulfasalazine, or antiepileptics if used for seizures (ok to use the latter if part of a pain regimen). Prior loperamide use for diarrhea is permitted at enrollment but should be changed to diphenoxylate / atropine before initiation of treatment.
* Has a history of psoriatic arthritis requiring systemic treatment.
* Has a history of porphyria.
* (Expansion phase only) Inability to safely undergo tumor biopsies (e.g. requirement for antiplatelet therapy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2019-10-22 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Up to 30 days
  Will employ the Bayesian optimal interval (BOIN) design to find the MTD.

SECONDARY OUTCOMES:
Response rate | Up to 1 year
Incidence of adverse events | Up to 1 year
  Toxicity will be assessed using common toxicity criteria version 5.
Progression free survival | Up to 1 year
  To determine the ability of the combination to halt tumor growth.
Overall survival | Up to 1 year
  To assess the overall survival of patients treated on this regimen.

OTHER OUTCOMES:
Somatic gene mutation profile | Up to 1 year
  Will be acquired by standard of care testing. Will compare the efficacy of treatment to somatic gene mutation profile.
Markers of autophagy | Up to 1 year
  Will assess pre- and post- treatment tissue to determine if markers of autophagy correlate with response to treatment.
Effect of this binimetinib/hydroxychloroquine treatment on changes in muscle and fat mass | Up to 1 year
  Will be analyzed by computed tomography scan (as standard of care treatment).

CONTACTS AND LOCATIONS:
Overall Officials: Shubham Pant, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org